CLINICAL TRIAL: NCT01718782
Title: Ventilation With Laryngeal Mask Ambu Aura Once vs. Supreme in Children
Brief Title: Laryngeal Mask Ambu Aura Once vs. Supreme in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Other studies with the same protocol have already published.
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Peter Paal, Peter Paal, MD, DESA, EDIC, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AN4111 292/4.23
Record Dates: First submitted 2012-09-27; First posted 2012-10-31 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Apnea
Keywords: laryngeal mask, leakage pressure, ventilation
MeSH Terms: conditions — Apnea; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laryngeal mask Ambu AuraOnce (Active Comparator): laryngeal mask Ambu AuraOnce
  Interventions: Device: laryngeal mask Ambu AuraOnce
- laryngeal mask LMA Supreme (Active Comparator): laryngeal mask LMA Supreme
  Interventions: Device: laryngeal mask LMA Supreme

INTERVENTIONS:
Device: laryngeal mask Ambu AuraOnce — airway management and mechanical ventilation with laryngeal mask
  Arms: laryngeal mask Ambu AuraOnce
Device: laryngeal mask LMA Supreme — airway management and mechanical ventilation with laryngeal mask
  Arms: laryngeal mask LMA Supreme

SUMMARY:
The purpose of this study is determine safety and efficiency of mechanical ventilation in children with two different types of single use laryngeal masks (Ambu AuraOnce vs. LMA Supreme). The main interest is leakage pressure of oropharynx and stomach. The null hypothesis is that leakage pressures of Ambu AuraOnce and LMA Supreme are equivalent. The alternative hypothesis is that there is a difference in leakage pressure.

DETAILED DESCRIPTION:
Before starting surgery patients will be anesthetised and airway managed either with LMA Ambu AuraOnce or Supreme. Ventilation parameters, stomach inflation, and hemodynamic parameters will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-10 years
* ASA I - III
* Elective procedure in general anaesthesia
* Parental informed consent

Exclusion Criteria:

* Non fasting patient
* Body mass index > 35 kg/m2
* Cervical spine pathologies or peripheral neurologic deficiences
* Malformations of upper airway or head
* Anamnestic hiatus hernia or esophageal reflux
* Status post operation of stomach or esophagus
* Recurrent respiratory infection or obstructive airway disease
* Non elective procedure

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Leakage pressure [cmH2O] | 1min
  After ventilation has been established the leakage pressure will be measured, ie 1min after establishing ventilation

SECONDARY OUTCOMES:
Efficient ventilation [mL], | 3min
  After ventilation has been established the efficient ventilation, tidal volume and stomach inflation will be measured, ie 3min after establishing ventilation
tidal volume [mL], | 3 minutes
stomach insufflation [yes or no] | 3 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Peter Paal, MD,DESA,EDIC, Principal Investigator — University Hospital Innsbruck, Department of Anaesthesia + Intensive Care
Locations (1):
- University Hospital Innsbruck, Innsbruck, Tyrol, Austria